CLINICAL TRIAL: NCT05699200
Title: Role of the Neurovascular System in Spontaneous Coronary Artery Dissection (SCAD)
Brief Title: A Study to Analyze the Role of Sympathetic Nervous System in Spontaneous Coronary Artery Dissection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marysia Tweet, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-005636; 1K23HL155506 (NIH)
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Spontaneous Coronary Artery Dissection; Healthy
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous | interventions — Echocardiography; Ultrasonography, Carotid Arteries; Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spontaneous coronary artery dissection (SCAD) group (Other): Subject with a history of SCAD will undergo a series of diagnostic studies to assess neurovascular function.
  Interventions: Other: Arterial Tonometry; Diagnostic Test: Echocardiogram; Diagnostic Test: Carotid Ultrasounds; Diagnostic Test: Elastography; Other: Ankle-Brachial Index; Other: Microneurography with sympathoexcitatory maneuvers
- Healthy Control Group (Other): Healthy subjects will undergo a series of diagnostic studies to assess neurovascular function.
  Interventions: Other: Arterial Tonometry; Diagnostic Test: Echocardiogram; Diagnostic Test: Carotid Ultrasounds; Diagnostic Test: Elastography; Other: Ankle-Brachial Index; Other: Microneurography with sympathoexcitatory maneuvers

INTERVENTIONS:
Other: Arterial Tonometry — We will measure arterial stiffness using arterial tonometry.
Diagnostic Test: Echocardiogram — We will collect limited ultrasound images of the heart.
Diagnostic Test: Carotid Ultrasounds — We will perform ultrasound imaging of the carotid artery.
Diagnostic Test: Elastography — We will measure the elastic properties of the arteries using elastography.
Other: Ankle-Brachial Index — We will measure the ankle-brachial index to assess peripheral artery blood flow.
Other: Microneurography with sympathoexcitatory maneuvers — We will measure sympathetic nerve activity at rest and in response to isometric handgrip, mental stress test, cold pressor test, Valsalva maneuvers.

SUMMARY:
The purpose of this research is to compare sympathetic function (flight or fight system) and arterial health including structure and mechanics of participants with history of spontaneous coronary artery dissection (SCAD) to age and sex matched control participants.

ELIGIBILITY:
Inclusion Criteria:

* For SCAD patients: history of SCAD as confirmed by coronary angiography or cardiac computed tomography angiography
* For controls: no cardiac disease history

Exclusion Criteria:

* Pregnancy
* Known or suspected unstable cardiac condition within 4 weeks of the study
* Active treatment with anticoagulation or dual antiplatelet therapy
* Prisoner

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Arterial thickness | Baseline
  Measured by carotid ultrasound intimal media thickness reporting in mm
Arterial stiffness | Baseline
  Measured by carotid ultrasound pulse wave velocity reporting in m/s
Baroreflex sensitivity | Baseline
  The slope between heart rate and blood pressure at rest and during the Valsalva Maneuver (ms/mmHg)
Sympathetic response to stress | Baseline
  Blood pressure or muscle sympathetic nerve activity response to sympathoexcitatory stressors (mm/Hg or bursts/min).

CONTACTS AND LOCATIONS:
Overall Officials: Marysia Tweet, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No